CLINICAL TRIAL: NCT00218426
Title: Addiction Treatment in Russia: Oral and Depot Naltrexone
Brief Title: Addiction Treatment in Russia: Oral vs. Naltrexone Implant
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-17317-1; R01DA017317 (NIH); R01-17317-1; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-02

CONDITIONS: Heroin Dependence; Opioid-Related Disorders
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ONP + DNI (Active Comparator): Oral naltrexone placebo (ONP) + Depot Naltrexone Implant (DNI) 1000 mg
  Interventions: Drug: naltrexone implant; Drug: oral placebo naltrexone
- ON + DNIP (Active Comparator): Oral naltrexone (ON) 50 mg + Depot Naltrexone placebo Implant (DNIP)
  Interventions: Drug: oral naltrexone; Drug: placebo implant
- ONP + DNIP (Placebo Comparator): Oral placebo naltrexone + placebo naltrexone implant
  Interventions: Drug: oral placebo naltrexone; Drug: placebo implant

INTERVENTIONS:
Drug: naltrexone implant — naltrexone implant is 1000 mg naltrexone
  Other Names: DNI
  Arms: ONP + DNI
Drug: oral naltrexone — oral naltrexone 50 mg/day
  Other Names: ON
  Arms: ON + DNIP
Drug: oral placebo naltrexone — oral placebo naltrexone resembles active medication
  Other Names: ONP
  Arms: ONP + DNI; ONP + DNIP
Drug: placebo implant — placebo implant resembles active medication
  Other Names: DNIP
  Arms: ON + DNIP; ONP + DNIP

SUMMARY:
Heroin addiction is a growing problem in Russia; individuals who enter heroin addiction treatment often relapse. Therefore, effective heroin addiction treatments are necessary to prevent relapse. The purpose of this study is to compare oral naltrexone with a naltrexone implant that provides opioid blockade for two months in preventing relapse to heroin addiction in St. Petersburg, Russia.

DETAILED DESCRIPTION:
The usual treatment of heroin addiction in Russia involves detoxification and 2-4 weeks of rehabilitation with referral to outpatient follow-up. Though most patients complete inpatient treatment, few keep follow-up appointments and relapse rates are high. More effective therapies are needed, especially in view of the epidemic of heroin addiction that has resulted in the spread of HIV and other infectious diseases. A recently-completed study of 52 patients randomized to oral naltrexone (ON) or oral naltrexone placebo (ONP) has shown efficacy in preventing relapse and reducing HIV risk but dropout was a problem with only 44% of ON patients proven to have not relapsed by 6 months (as compared to 16% of ONP patients). A larger study of 280 patients randomized to ON or ONP replicated these results and found some indication that adding an selective serotonin reuptake inhibitor (SSRI) to naltrexone may improve its efficacy in women, probably because they tend to have higher levels of psychiatric symptoms than men.

We think that retention and outcome can be improved by using a longer acting naltrexone preparation, and in this study we propose to compare ON with a depot naltrexone implant (DNI) that is manufactured and approved for use in Russia, and provides opioid blockade for 8-10 weeks. We will use a placebo-controlled, double-blind/double-dummy design since a placebo-controlled trial is required by the Russian equivalent of our FDA as a condition for testing a pharmacotherapy. Participants will be male and female heroin addicts who have been detoxified in addiction treatment hospitals or outpatient settings in St. Petersburg and have a family member willing and able to supervise medication adherence and facilitate follow-up. After giving informed consent and confirming the absence of physiologic dependence, 306 patients will be randomly assigned to a 6-month treatment in one of three groups of 102 each: oral naltrexone (ON) + depot naltrexone implant placebo (DNIP); oral naltrexone placebo (ONP) + depot naltrexone implant (DNI); or ONP + DNIP. All patients will receive biweekly clinical management/adherence enhancement counseling. Assessments will be done at baseline, at each biweekly appointment during the 6-months of medication treatment, and at 3 and 6 months following the end of study medication. Primary outcome will be the relapse free proportion at months 1-6; secondary outcomes will be time to dropout, opioid positive urines, HIV risk, use of alcohol and other drugs, psychiatric symptoms, and other measures of overall adjustment. We hypothesize that outcomes will be better with DNI than ON, and that each will be more effective than placebo.

ELIGIBILITY:
Inclusion Criteria:

* Current opioid dependence
* Recently completed opioid detoxification

Exclusion Criteria:

* Serious medical or psychiatric condition requiring immediate hospitalization or that would make participation in the study hazardous
* Planning to leave the study area within the 12 months following study entry
* Imminent incarceration
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 306 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2010-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Woody, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States
- Pavlov Medical University, Saint Petersburg, Russia

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- [Derived] Krupitsky E, Zvartau E, Blokhina E, Verbitskaya E, Wahlgren V, Tsoy-Podosenin M, Bushara N, Burakov A, Masalov D, Romanova T, Tyurina A, Palatkin V, Yaroslavtseva T, Pecoraro A, Woody G. Anhedonia, depression, anxiety, and craving in opiate dependent patients stabilized on oral naltrexone or an extended release naltrexone implant. Am J Drug Alcohol Abuse. 2016 Sep;42(5):614-620. doi: 10.1080/00952990.2016.1197231. Epub 2016 Jul 19. PMID 27436632

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects (SS) are from Leningrad Regional Alcoholism and Substance Abuse Treatment Center, Leningrad Region; and St. Petersburg City Alcoholism and Substance Abuse Treatment Center, screened for detoxification and if met study criteria and interested were referred to study on day of discharge. First SS admitted on 7/31/06, last visit was 1/4/09.
Pre-assignment Details: SS were opioid dependent with physiological features for at least 1 year, negative urine for opioids, had ability to give informed consent, not on psychotropic medication, if female, not pregnant, could provide at least 1 relative contact, no significant lab abnormality, and not major psych disorder.
Groups:
- ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant: Oral naltrexone
  Oral naltrexone: oral naltrexone 50 mg/day
  DNIP
  Depot Placebo Naltrexone Implant
- DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo: naltrexone implant
  naltrexone implant: The implant is 1000 mg naltrexone
  ONP oral naltrexone placebo tablet
- ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant: ONP daily placebo oral naltrexone
  monthly placebo depot naltrexone implant
Period: Overall Study
Arm/Group | ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant | DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo | ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant
Started | 102 | 102 | 102
Completed | 54 | 16 | 11
Not Completed | 48 | 86 | 91

BASELINE CHARACTERISTICS:
Groups:
- ONP + DNI: Oral naltrexone placebo + Depot Naltrexone Implant 1000 mg
  naltrexone implant: depot implant is 1000 mg naltrexone
  placebo oral tablet: placebo oral tablet resembles active medication
- ON + DNIP: Oral naltrexone 50 mg + Depot Naltrexone placebo Implant
  oral naltrexone: oral naltrexone 50 mg/day
  depot placebo implant: placebo implant resembles active medication
- ONP + DNIP: Oral placebo naltrexone + placebo naltrexone implant
  placebo oral tablet: placebo oral tablet resembles active medication
  depot placebo implant: placebo implant resembles active medication
- Total: Total of all reporting groups
Arm/Group | ONP + DNI | ON + DNIP | ONP + DNIP | Total
Number analyzed (Participants) | 102 | 102 | 102 | 306
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 102 | 102 | 102 | 306
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 28.0 [18 to 40] | 27.9 [18 to 40] | 28.7 [18 to 40] | 28.2 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 28 | 84
  Male | 74 | 74 | 74 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 102 | 102 | 102 | 306
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 102 | 102 | 102 | 306
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 102 | 102 | 102 | 360

OUTCOME MEASURES:

1. Primary Outcome: Retention Without Relapse to Heroin Addiction (Measured at Month 6)
Description: Survival analysis (Kaplan-Meier survival functions with log-rank Cox-Mantel criteria for group comparison was used to determine the primary outcome of retention, defined as not missing 2 consecutive counseling sessions and not having a relapse. Because this outcome combined patients who failed to keep appointments with those who kept appointments but relapsed, the proportion of non-survivors attributable to proven relapse.
Time Frame: 6 months
Population: Subjects who remained in treatment without relapse. remaining in treatment = 6 months manualized clinical counseling, plus medication.
Measure: Count of Participants; unit: Participants
Arm/Group | ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant | DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo | ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant
Number analyzed (Participants) | 102 | 102 | 102
Participants | 54 | 16 | 11

2. Secondary Outcome: Number of Subjects Who Dropped Out of Treatment
Description: Kaplan-Meier survival curves for the event of subjects who dropped out of treatment
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant | DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo | ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant
Number analyzed (Participants) | 102 | 102 | 102
participants | 54 | 16 | 11

3. Secondary Outcome: Positive Opioid Urine Test
Description: missed urine tests were imputed to be positive for opiates
Time Frame: 6 months
Population: missing = positive; results negative for opioids
Measure: Number (95% Confidence Interval); unit: urine tests
Units Other Than Participants: urine tests
Arm/Group | ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant | DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo | ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant
Number analyzed (Participants) | 102 | 102 | 102
Number analyzed (urine tests) | 1428 | 1428 | 1428
urine tests | .427 [0.40 to 0.45] | .636 [0.60 to 0.66] | .341 [0.32 to 0.37]

4. Secondary Outcome: Use of Alcohol
Description: use of alcohol grams per day
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant | DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo | ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant
Number analyzed (Participants) | 102 | 102 | 102
grams per day | 10.2 (1.7) | 9.0 (1.7) | 9.6 (1.6)

5. Secondary Outcome: Composite Score of Psychiatric Problems
Description: composite score is a decimal score; with 0 = no problems, 1 = the most problems based on the Addiction Severity Index composite score of 11 indexed questions.
Time Frame: 6 months
Population: mean of composite score
Measure: Mean (Standard Deviation); unit: composite score
Arm/Group | ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant | DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo | ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant
Number analyzed (Participants) | 102 | 102 | 102
composite score | 0.19 (0.02) | 0.15 (0.02) | 0.18 (0.02)

6. Secondary Outcome: HIV Risk (Baseline)
Description: The Risk Assessment Behavior (RAB), is an HIV risk Scale. The Total Score is scored by adding the values that correspond to the responses selected by the subject for the items asked. This highest total score is 40 (highest risk), and the lowest score = 0 (no risk). This assessment has 2 Subsections: 1) Drug Risk = 8 questions (lowest Drug Risk score = 0 (no risk), and highest drug risk score = 22 =(greatest risk), 2) 10 Sex Risk questions: scores are 0 = no risk, and 18 = highest risk). Total RAB Score = Drug Risk Total + Sex Risk Total (0 = no risk, 40 = highest). See: Risk Assessment Battery (RAB) Scoring System, https://www.med.upenn.edu/hiv/assets/user-content/.../RABScoringv2.112.21.95.doc
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant | DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo | ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant
Number analyzed (Participants) | 102 | 102 | 102
score on a scale | 8.1 (0.44) | 8.0 (0.47) | 8.7 (0.49)

7. Secondary Outcome: Global Assessment Form (GAF)
Description: Assessment of overall psychiatric function comprises Axis V in the DSM-IV (DSM-IV, 1994). GAF scores range from 0 to 100. A reasonably well-functioning person will score above 70; serious impairment is below 50.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant | DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo | ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant
Number analyzed (Participants) | 102 | 102 | 102
score on a scale | 62.8 (0.7) | 64.7 (0.8) | 62.5 (0.9)

8. Secondary Outcome: Amphetamine Drug Use
Description: Number of subjects who used Amphetamine in the past 90 days at baseline as measured by the TimeLine Follow-back Form (TLFB) . The TLFB is an instrument that assesses substance use over a specified period of time (Sobel & Sobel, 1992).
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant | DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo | ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant
Number analyzed (Participants) | 102 | 102 | 102
Participants | 6 | 12 | 18

9. Secondary Outcome: Cocaine Drug Use
Description: Number of subjects with cocaine drug use in the past 90 days at baseline as measured by the TimeLine Follow-back Form (TLFB) . The TLFB is an instrument that assesses substance use over a specified period of time (Sobel & Sobel, 1992).
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ONP + DNI | ON + DNIP | ONP + DNIP
Number analyzed (Participants) | 102 | 102 | 102
Participants | 0 | 0 | 0

10. Secondary Outcome: Marijuana Drug Use
Description: Number of subjects with Marijuana use in the past 90 days at baseline as measured by the TimeLine Follow-back Form (TLFB) . The TLFB is an instrument that assesses substance use over a specified period of time (Sobel & Sobel, 1992).
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant | DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo | ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant
Number analyzed (Participants) | 102 | 102 | 102
Participants | 22 | 35 | 25

11. Secondary Outcome: Benzodiazepine Drug Use
Description: Number of subjects with benzodiazepine drug use in the past 90 days at baseline as measured by the TimeLine Follow-back Form (TLFB) . The TLFB is an instrument that assesses substance use over a specified period of time (Sobel & Sobel, 1992).
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant | DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo | ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant
Number analyzed (Participants) | 102 | 102 | 102
Participants | 10 | 15 | 9

ADVERSE EVENTS:
Time Frame: 3 Years
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product. The event need not have a causal relationship to the treatment. Normal withdrawal is not considered an adverse event.
Arm/Group | ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant | DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo | ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/102 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/102 | 1/102
Other Adverse Events (participants affected / at risk) | 6/102 | 17/102 | 3/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant (N=102) | DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo (N=102) | ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant (N=102)
cholecystectomy (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ON + DNIP, Oral Naltrexone + Depot Placebo Naltrexone Implant (N=102) | DNI + ONP , Naltrexone Implant + Oral Naltrexone Placebo (N=102) | ONP + DNIP, Oral Placebo Naltrexone and Depot Placebo Implant (N=102)
headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
drowsiness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
high blood pressure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0)
increased liver enzyme (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
local site reaction (Surgical and medical procedures) | 2 (2) | 9 (9) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations include limited amount of data on patients who did not remain in treatment, thus making it difficult to obtain more accurate information on the proportions with relapse at 9- and 12- month follow-ups and other secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No